CLINICAL TRIAL: NCT00626938
Title: Proteomics as a Tool for Biomarker Detection in Sarcoidosis
Brief Title: Role of Proteomics in Diagnosing Sarcoidosis
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, marjolein drent, Prof. Marjolein Drent, Maastricht University Medical Center
Other Study IDs: MEC 04-145.11
Record Dates: First submitted 2008-02-14; First posted 2008-02-29 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Sarcoidosis
Keywords: sarcoidosis; protein profile; CYP-450; TNF-alpha polymorphisms; HLA
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood will be collected from all participants, but all samples will be stored anonymously.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- sarcoidosis: sarcoidosis patients
- controls: healthy volunteers and other interstitial lung disease (ILD) patients

SUMMARY:
Sarcoidosis is a multi-systemic disorder, meaning that it can involve any organ in the body and that its clinical presentation is highly variable. In 90% of all sarcoidosis cases the lungs are affected. It is difficult to give a concise definition of sarcoidosis due to the fact that its exact cause is still unknown. Consequently, diagnosing the disease is also rather difficult. Up till now, sarcoidosis is generally diagnosed by using general clinical methods to evaluate the status of the lung including a chest X-ray, lung biopsy and bronchoalveolar lavage (BAL). However, some of these methods are considered to be rather invasive and, even more important, non-conclusive. Therefore, the current study has been designed to evaluate the use of a new technique, called SELDI-TOF mass spectrophotometry, for the diagnosis of sarcoidosis. This technique enables the analysis of all enzymes present in the blood of sarcoidosis patients which may hopefully lead to creating a disease-specific protein-profile that may facilitate the recognition of sarcoidosis. Moreover, these results will be compared with other currently used laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pulmonary sarcoidosis stage I-IV

Exclusion Criteria:

* Non-smoking
* No treatment for extra-pulmonary symptoms of sarcoidosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting the out-patient clinic of the university hospital Maastricht.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2005-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
protein profile in blood | within 1 month after obtaining sample

SECONDARY OUTCOMES:
CYP and TNF polymorphisms | within 6 months after obtaining sample

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein Drent, Prof,MD,PhD, Study Director — University Hospital Maastricht, Departement of Respiratory Medicine; Otto Bekers, PhD, Principal Investigator — University Hospital Maastricht, Departement of Clinical Chemistry; Christine Voorter, PhD, Principal Investigator — University Hospital Maastricht, Departement of Tissue Typing; Marja P van Dieijen-Visser, Prof,MSc,PhD, Study Chair — University Hospital Maastricht, Departement of Clinical Chemistry
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands